CLINICAL TRIAL: NCT05263661
Title: Ligation of Intersphincteric Fistula Tract Versus Rectal Advancement Flap in the Treatment of Complex Anal Fistula: Randomised Clinical Trial
Brief Title: Ligation of Intersphincteric Fistula Tract Versus Rectal Advancement Flap in the Treatment of Complex Anal Fistula
Acronym: LIFTRAF-RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital General Universitario Reina Sofía de Murcia (Other)
Responsible Party: Principal Investigator, Jorge Alejandro Benavides Buleje, Principal Investigator, Hospital General Universitario Reina Sofía de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIFTRAF-RCT; JBB1 (Other: HGU Reina Sofia's CEIC)
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anal Fistula
Keywords: anal fistula, lift, advancement flap, recurrence
MeSH Terms: conditions — Rectal Fistula; Recurrence

STUDY DESIGN:
Intervention Model Description: A controlled, randomised clinical trial
Who Masked: Outcomes Assessor
Masking Description: Open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFT (Experimental): ligation of interesphincteric fistula tract
  Interventions: Procedure: LIFT
- FLAP (Active Comparator): Rectal advancement flap
  Interventions: Procedure: FLAP

INTERVENTIONS:
Procedure: LIFT — Ligation of fistula tract between external and internal sphincter
  Other Names: ligation of interesphincteric fistula tract
  Arms: LIFT
Procedure: FLAP — Creation of a partial wall rectal flap to close internal opening of fistula tract
  Other Names: Rectal advancement flap
  Arms: FLAP

SUMMARY:
Objective: Rectal advancement flap (RAF) is currently considered the gold standard in the treatment of complex anal fistula (CAF). Clinical trials are a priority given the few consistent results available with level 1 evidence. We compare the results of two conservative sphincter techniques: ligation of intersphincteric fistula tract (LIFT) versus RAF.

Material and Method: A controlled, randomised clinical trial is conducted in patients operated between 2013 and 2016 in Hospital General Universitario Reina Sofia, Murcia, Spain. The primary objective was to evaluate relapse at 12 months of follow-up, and the secondary objectives were post-op anal continence (Wexner), post-operative complications (haematoma, infection of surgical site, suture dehiscence), duration of surgery and hospitalisation. Post-operative controls 1, 3, 6 and 12 months after surgery.

DETAILED DESCRIPTION:
Material and method

Design:

Phase III, single centre, randomised, open-label, parallel group trial controlled with active comparator, with blind evaluation of results by a non-commercial third party. This study was conducted in 72 patients who had undergone complex anal fistula surgery and met the inclusion criteria.

The study was conducted by the Colo proctology Unit of the General and Digestive Surgery Department of Hospital General Universitario Reina Sofia, Murcia, Spain, from February 2013 to June 2016, and approved by the hospital's Independent Ethics Committee (IEC). The study was conducted pursuant to the principles of the Declaration of Helsinki (Seoul, October 2008) and the Good Clinical Practice (GP) standards of the European Economic Community's task force on the efficacy of medicinal substances (1990) and all legislation currently applicable in Spain (Royal Decree 223/2004 of 6 February).

Patients with a diagnosis or suspected diagnosis of anal fistula were referred to the Coloproctology Office. At the first visit, demographic data and a clinical history was obtained, followed by a physical examination of the anal region, with rigid anoscopy, ordering an endoanal ultrasound. At a second visit, if the diagnosis of complex anal fistula was confirmed, after providing information about the study, the patient was invited to participate, signed the consent form, and underwent the pre-operative Wexner scale. Patients were allocated a randomisation code for LIFT or RAF on the day of surgery. After surgery, controls were performed on days 7 and 14, by means of a symptoms diary to be completed by each patient, and 1, 3, 6 and 12 months after the surgery, with the Wexner scale calculated in the last control of each patient.

Complex anal fistula was defined as a fistula at risk of affecting continence involving more than 30% of the sphincteric apparatus. Infection of surgical site at or near the incision in the 30 days following surgery (28). Haematoma was defined as accumulation of blood in the surgical area, with bluish or violet colouring of the affected area; surgical wound dehiscence was defined as the spontaneous separation of the edges of the wound, in the absence of surgical site infection.

The inclusion criteria were patient diagnosed with transsphincteric (medium or high) or suprasphincteric cryptoglandular anal fistula, over 18 years of age, with no abscess at the time of surgery, who agreed to participate and signed the informed consent form, and was capable transsphincteric understanding and following study instructions. The exclusion criteria were minor patient, diagnosed with, or with a suspected diagnosis of, Crohn's disease, malignant anal tumour, tuberculosis or suppurative hidradenitis, a history of radiotherapy of the ano-perineal region, language difficulties that prevent comprehension of the study, or refusal to participate.

Each patient's data were collected in the case report form and transferred to a database for their statistical analysis by an analyst unrelated to the study, preserving their anonymity and the treatment group to which they belonged.

Study objectives:

The primary objective was to show the non-inferiority in therapeutic efficacy of LIFT versus RAF in the surgical treatment of CAF. The primary efficacy endpoint was the proportion of subjects in each treatment group without fistula recurrence 12 months after surgery.

The secondary objectives were to show the non inferiority of LIFT versus RAF in therapeutic safety:

* Evaluating functionality, both before and after surgery, in both treatment groups, through anal continence, using the Wexner scale.
* Comparing post-operative complications in both treatment groups: infection of surgical site, haematoma and surgical wound dehiscence.
* Comparing time to fistula relapse in both treatment groups, by a survival analysis.
* Analysing hospital management factors (duration of surgery and hospitalisation) in both treatment groups.

Randomisation and surgeries:

The subjects were randomised 1:1 to receive LIFT or RAF surgery. Patient randomisation was by randomisation in balanced six-cell blocks; the sequence was custodied by the Teaching Secretary, unrelated to the study. The surgeon requested each patient's randomisation code on the day of surgery. LIFT or RAF.

The patients were operated by three surgeons from the Coloproctology Unit, whose learning curve was based on unifying experimental technique (LIFT) criteria in six patients before the start of the study. All the surgeries used epidural anaesthesia.

* Ligation of the intersphincteric fistula tract (LIFT): jackknife position. Location of IFO by injecting a diluted (1/3) solution of hydrogen peroxide through the external fistula orifice (EFO). Opening of the fistula trajectory with a stylus. Curved 2.5 cm incision in the intersphincteric space until trajectory is skeletalised, ligation of internal and external sphincter with 3/0 single thread polyglecaprone 25 absorbable suture (MonocrylTM Plus®), exeresis of the trajectory between the ligations with cold scalpel. Cleansing of distal part with curette and enlargement of the external fistula orifice (EFO). Closure of the muscular intersphincteric plane with loose stitches of 3/0 polyglecaprone 25 single-thread absorbable suture (MonocrylTM Plus®). Closure of intersphincteric skin with simple plaited polyglycolic acid absorbable sutures (SSA90®).
* Rectal advancement flap (CAR): jackknife in case of anterior fistula and lithotomy in case of posterior fistula. Location of IFO by injecting a diluted (1/3) solution of hydrogen peroxide through EFO. Opening of the fistula trajectory with a stylus. Excision of the extrasphincteric component of the fistula and cleansing of sphincteric tract. Design of a flap with electric scalpel, of partial thickness including mucosa-submucosa and part of the fibres of the internal sphincter, with a broad base (twice the apex), sliding in a craniocaudal direction, without tension, to completely cover the internal part of the fistula, closure of the internal orifice with cross stitch and suture of flap with simple 3/0 polyglecaprone 25 absorbable suture (MonocrylTM Plus®).

Peri-operative care and follow-up:

All patients were advised to follow a waste-free diet 48 hours before admission, and were given an enema on the night before surgery. All patients received antibiotic prophylaxis with IV amoxicillin/clavulanic acid 2 g half an hour before the start of surgery. Six hours after surgery, liquid diet commenced, progressing to semi-bland for dinner that night, and bland on the first day after surgery. No postoperative antibiotic treatment was indicated. The ward surgeon, unrelated to the study, discharged the patient based on these criteria: afebrile, controlled pain, appropriate oral tolerance and surgical wound correct.

All patients received 12 months of follow-up, except for one who left the study after 8 months. After discharge, the patient attended for cleaning of the surgical wound on the following two Fridays, with review of the symptom diary (SD) and evaluation of possible complications by the Coloproctology Unit surgeon. The patient attended a scheduled appointment one month after surgery (1st post-op visit), where he was evaluated and data was collected in the case report form (CRF), the SD was collected and possible complications were evaluated (infection of surgical site, haematoma, wound dehiscence). New appointments were scheduled at 3 (2nd post-op visit) and 6 months (3rd post-op visit), where the patient was evaluated and the respective data were collected. The final visit (4th post-op visit) took place at 12 months, where the post-op Wexner scale was applied.

Sample size and statistical analysis:

When the study began, publications reported a relapse rate of 0-33% with rectal advancement flap, with an average of 19% (19) and we can assume that the response rate to surgical treatment was approximately 85% for RAF, while the expected response rate for LIFT was 70%, the average of the rates observed in clinical studies published to date, which ranged from 57% to 94% (19).

With these data, considering response as the absence of fistula recurrence at 12 months, and in order to obtain a power of 80% to reject the null hypothesis (Ho), that the difference between proportions p1 and p2 was lower than the non-inferiority limit, by a normal asymptotic test for proportions, unilateral for two independent samples, considering that the level of significance was 0.5, assuming that the proportion in the reference group was 85%, the proportion in the experimental group was 70%, the proportion of patients in the reference group relative to the total was 50% and the non-inferiority limit was 10% and the expected withdrawal rate was 5%, 36 patients were required for the reference group and 36 for the experimental group, making a total of 72 patients in the study.

The categorical variables were described with mean values and percentages. The continuous variables were described with mean values and standard deviation, or median values and range. The Chi-square or Fisher test was used to compare two qualitative variables, to see whether there was dependence between them. The Bonferroni correction was used for column comparisons. The Student's t-test was used for comparison of the two groups, after checking the normality and homogeneity of variances assumptions with the Kolmogorov-Smirnov and Levene tests, respectively. For the analysis of non-inferiority of the primary and categorical variables, the calculation was through the Farrington-Manning score and Miettinen-Nurminen Score tests, with a level of significance of 0.05 and a non-inferiority limit of 0.10. For the continuous variables, non-inferiority was evaluated by difference of means, with the Mann-Whitney U-test and the Wilcoxon test. All statistical comparisons used a bilateral test with a level of significance of p < 0.05.

The primary study analysis was based on the intention-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with transsphincteric (medium or high) or suprasphincteric cryptoglandular anal fistula
* with no abscess at the time of surgery
* who agreed to participate and signed the informed consent form
* capable transsphincteric understanding and following study instructions

Exclusion Criteria:

* diagnosed with, or with a suspected diagnosis of, Crohn's disease
* diagnosed with, or with a suspected diagnosis of, malignant anal tumour
* diagnosed with, or with a suspected diagnosis of,tuberculosis or suppurative hidradenitis
* a history of radiotherapy of the ano-perineal region
* language difficulties that prevent comprehension of the study
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Curation | 1 year
  Proportion of subjects in each treatment group without fistula recurrence after surgery

SECONDARY OUTCOMES:
Functionality | 1 year
  Anal continence measured by Wexner Scale (0-20, higher is worst)
Security | 1 month
  Rate of Complications after surgery
Time of recurrence | 10 years
  time to fistula relapse afeter surgery
Time of surgery | 1 day
  Duration of surgery in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alejandro Benavides Buleje, PhD, Principal Investigator — Hospital General Universitario Reina Sofía

IPD SHARING:
Plan to Share IPD: No
If asked

REFERENCES:
- [Background] Sahnan K, Askari A, Adegbola SO, Tozer PJ, Phillips RKS, Hart A, Faiz OD. Natural history of anorectal sepsis. Br J Surg. 2017 Dec;104(13):1857-1865. doi: 10.1002/bjs.10614. Epub 2017 Aug 31. PMID 28857130
- [Background] Parks AG, Gordon PH, Hardcastle JD. A classification of fistula-in-ano. Br J Surg. 1976 Jan;63(1):1-12. doi: 10.1002/bjs.1800630102. PMID 1267867
- [Background] Sneider EB, Maykel JA. Diagnosis and management of symptomatic hemorrhoids. Surg Clin North Am. 2010 Feb;90(1):17-32, Table of Contents. doi: 10.1016/j.suc.2009.10.005. PMID 20109630
- [Result] Bleier JI, Moloo H. Current management of cryptoglandular fistula-in-ano. World J Gastroenterol. 2011 Jul 28;17(28):3286-91. doi: 10.3748/wjg.v17.i28.3286. PMID 21876615
- [Result] Cadeddu F, Salis F, Lisi G, Ciangola I, Milito G. Complex anal fistula remains a challenge for colorectal surgeon. Int J Colorectal Dis. 2015 May;30(5):595-603. doi: 10.1007/s00384-014-2104-7. Epub 2015 Jan 9. PMID 25566951
- [Result] Narang SK, Keogh K, Alam NN, Pathak S, Daniels IR, Smart NJ. A systematic review of new treatments for cryptoglandular fistula in ano. Surgeon. 2017 Feb;15(1):30-39. doi: 10.1016/j.surge.2016.02.002. Epub 2016 Mar 15. PMID 26993759
- [Result] Bubbers EJ, Cologne KG. Management of Complex Anal Fistulas. Clin Colon Rectal Surg. 2016 Mar;29(1):43-9. doi: 10.1055/s-0035-1570392. PMID 26929751
- [Result] Phillips J, Lees N, Arnall F. Current management of fistula-in-ano. Br J Hosp Med (Lond). 2015 Mar;76(3):142, 144-7. doi: 10.12968/hmed.2015.76.3.142. PMID 25761803
- [Result] Jacob TJ, Perakath B, Keighley MR. Surgical intervention for anorectal fistula. Cochrane Database Syst Rev. 2010 May 12;(5):CD006319. doi: 10.1002/14651858.CD006319.pub2. PMID 20464741
- [Result] Sandborn WJ, Fazio VW, Feagan BG, Hanauer SB; American Gastroenterological Association Clinical Practice Committee. AGA technical review on perianal Crohn's disease. Gastroenterology. 2003 Nov;125(5):1508-30. doi: 10.1016/j.gastro.2003.08.025. No abstract available. PMID 14598268
- [Result] de Groof EJ, Cabral VN, Buskens CJ, Morton DG, Hahnloser D, Bemelman WA; research committee of the European Society of Coloproctology. Systematic review of evidence and consensus on perianal fistula: an analysis of national and international guidelines. Colorectal Dis. 2016 Apr;18(4):O119-34. doi: 10.1111/codi.13286. PMID 26847796
- [Result] Jarrar A, Church J. Advancement flap repair: a good option for complex anorectal fistulas. Dis Colon Rectum. 2011 Dec;54(12):1537-41. doi: 10.1097/DCR.0b013e31822d7ddd. PMID 22067182
- [Result] Gottgens KW, Smeets RR, Stassen LP, Beets G, Breukink SO. Systematic review and meta-analysis of surgical interventions for high cryptoglandular perianal fistula. Int J Colorectal Dis. 2015 May;30(5):583-93. doi: 10.1007/s00384-014-2091-8. Epub 2014 Dec 10. PMID 25487858
- [Result] Rojanasakul A, Pattanaarun J, Sahakitrungruang C, Tantiphlachiva K. Total anal sphincter saving technique for fistula-in-ano; the ligation of intersphincteric fistula tract. J Med Assoc Thai. 2007 Mar;90(3):581-6. PMID 17427539
- [Result] Matos D, Lunniss PJ, Phillips RK. Total sphincter conservation in high fistula in ano: results of a new approach. Br J Surg. 1993 Jun;80(6):802-4. doi: 10.1002/bjs.1800800651. PMID 8330181
- [Result] Bleier JI, Moloo H, Goldberg SM. Ligation of the intersphincteric fistula tract: an effective new technique for complex fistulas. Dis Colon Rectum. 2010 Jan;53(1):43-6. doi: 10.1007/DCR.0b013e3181bb869f. PMID 20010349
- [Result] Balciscueta Z, Uribe N, Balciscueta I, Andreu-Ballester JC, Garcia-Granero E. Rectal advancement flap for the treatment of complex cryptoglandular anal fistulas: a systematic review and meta-analysis. Int J Colorectal Dis. 2017 May;32(5):599-609. doi: 10.1007/s00384-017-2779-7. Epub 2017 Feb 28. PMID 28247060
- [Result] Garg P. Randomized clinical trial of anal fistula plug versus endorectal advancement flap for the treatment of high cryptoglandular fistula in ano (Br J Surg 2009; 96: 608-612). Br J Surg. 2009 Aug;96(8):958-9; author reply 959. doi: 10.1002/bjs.6772. No abstract available. PMID 19591140
- [Result] Bondi J, Avdagic J, Karlbom U, Hallbook O, Kalman D, Saltyte Benth J, Naimy N, Oresland T. Randomized clinical trial comparing collagen plug and advancement flap for trans-sphincteric anal fistula. Br J Surg. 2017 Aug;104(9):1160-1166. doi: 10.1002/bjs.10549. Epub 2017 May 10. PMID 28489253
- [Result] Malakorn S, Sammour T, Khomvilai S, Chowchankit I, Gunarasa S, Kanjanasilp P, Thiptanakij C, Rojanasakul A. Ligation of Intersphincteric Fistula Tract for Fistula in Ano: Lessons Learned From a Decade of Experience. Dis Colon Rectum. 2017 Oct;60(10):1065-1070. doi: 10.1097/DCR.0000000000000880. PMID 28891850
- [Result] Xu Y, Tang W. Ligation of Intersphincteric Fistula Tract Is Suitable for Recurrent Anal Fistulas from Follow-Up of 16 Months. Biomed Res Int. 2017;2017:3152424. doi: 10.1155/2017/3152424. Epub 2017 Feb 8. PMID 28271064
- [Result] Mushaya C, Bartlett L, Schulze B, Ho YH. Ligation of intersphincteric fistula tract compared with advancement flap for complex anorectal fistulas requiring initial seton drainage. Am J Surg. 2012 Sep;204(3):283-9. doi: 10.1016/j.amjsurg.2011.10.025. Epub 2012 May 19. PMID 22609079
- [Result] Madbouly KM, El Shazly W, Abbas KS, Hussein AM. Ligation of intersphincteric fistula tract versus mucosal advancement flap in patients with high transsphincteric fistula-in-ano: a prospective randomized trial. Dis Colon Rectum. 2014 Oct;57(10):1202-8. doi: 10.1097/DCR.0000000000000194. PMID 25203377
- [Result] Roig JV, Jordan J, Garcia-Armengol J, Esclapez P, Solana A. Changes in anorectal morphologic and functional parameters after fistula-in-ano surgery. Dis Colon Rectum. 2009 Aug;52(8):1462-9. doi: 10.1007/DCR.0b013e3181a80e24. PMID 19617761
- [Result] Ye F, Tang C, Wang D, Zheng S. Early experience with the modificated approach of ligation of the intersphincteric fistula tract for high transsphincteric fistula. World J Surg. 2015 Apr;39(4):1059-65. doi: 10.1007/s00268-014-2888-1. PMID 25472892
- [Result] Sirikurnpiboon S, Awapittaya B, Jivapaisarnpong P. Ligation of intersphincteric fistula tract and its modification: Results from treatment of complex fistula. World J Gastrointest Surg. 2013 Apr 27;5(4):123-8. doi: 10.4240/wjgs.v5.i4.123. PMID 23671739
- [Result] Yassin NA, Hammond TM, Lunniss PJ, Phillips RK. Ligation of the intersphincteric fistula tract in the management of anal fistula. A systematic review. Colorectal Dis. 2013 May;15(5):527-35. doi: 10.1111/codi.12224. PMID 23551996
- [Result] Vergara-Fernandez O, Espino-Urbina LA. Ligation of intersphincteric fistula tract: what is the evidence in a review? World J Gastroenterol. 2013 Oct 28;19(40):6805-13. doi: 10.3748/wjg.v19.i40.6805. PMID 24187455
- [Result] Williams G, Williams A, Tozer P, Phillips R, Ahmad A, Jayne D, Maxwell-Armstrong C. The treatment of anal fistula: second ACPGBI Position Statement - 2018. Colorectal Dis. 2018 Jul;20 Suppl 3:5-31. doi: 10.1111/codi.14054. PMID 30178915
- [Result] Gecse KB, Bemelman W, Kamm MA, Stoker J, Khanna R, Ng SC, Panes J, van Assche G, Liu Z, Hart A, Levesque BG, D'Haens G; World Gastroenterology Organization, International Organisation for Inflammatory Bowel Diseases IOIBD, European Society of Coloproctology and Robarts Clinical Trials; World Gastroenterology Organization International Organisation for Inflammatory Bowel Diseases IOIBD European Society of Coloproctology and Robarts Clinical Trials. A global consensus on the classification, diagnosis and multidisciplinary treatment of perianal fistulising Crohn's disease. Gut. 2014 Sep;63(9):1381-92. doi: 10.1136/gutjnl-2013-306709. Epub 2014 Jun 20. PMID 24951257